CLINICAL TRIAL: NCT02986360
Title: Informed Implementation of Breast Density Reporting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jennifer S. Haas, MD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016P001411
Record Dates: First submitted 2016-09-12; First posted 2016-12-08 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Breast Density, Breast Cancer Prevention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vidscrip educational video (Active Comparator): Patients receive Vidscrip education video discussing breast density in the context of their normal mammogram result
  Interventions: Behavioral: Vidscrip educational video
- Standard of care (No Intervention): Receive normal mammogram result and standard letter about breast density without any additional educational tools to contextualize breast density

INTERVENTIONS:
Behavioral: Vidscrip educational video — Vidscrip educational video provide to women
  Arms: Vidscrip educational video

SUMMARY:
1. To develop brief informational videos, Vidscrips, that can be sent to women following their mammogram to provide personalized information that integrates breast density with overall breast cancer risk, and provides information about additional care recommendations and talking tips for conversations with the health care providers.
2. To test the effectiveness of this tool in a trial of 300 women undergoing mammography. The investigators hypothesize that individuals in the intervention arm (vs. those in the standard care arm who receive a letter with the language required by the legislation) will have more accurate knowledge of their overall risk of breast cancer, their Mammographic Breast Density (MBD) result, more appropriate observed and intended use of additional screening [i.e., use of screening Magnetic Resonance Imaging (MRI) will be reserved only for women at high risk of breast cancer], better satisfaction with their episode of breast cancer screening, less decisional conflict about their personal decision for any additional evaluation, and less worry about breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* undergoing screening mammography at participating hospital facility
* normal mammogram result
* no prior history of Ductal carcinoma in situ (DCIS) or invasive breast cancer
* must have email account

Exclusion Criteria:

* non-English speaking
* prior history of Ductal Carcinoma in situ (DCIS) or invasive breast cancer
* no email

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Knowledge of overall breast cancer risk | 1 month
  electronic questionnaire developed by research staff
Knowledge of breast density | 1 month
  electronic questionnaire developed by research staff

SECONDARY OUTCOMES:
Observed use of additional screening | 9 months of index mammogram
  Additional screening tests (ultrasound or MRI) extracted from patient's electronic medical record

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer S Haas, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haas JS, Giess CS, Harris KA, Ansolabehere J, Kaplan CP. Randomized Trial of Personalized Breast Density and Breast Cancer Risk Notification. J Gen Intern Med. 2019 Apr;34(4):591-597. doi: 10.1007/s11606-018-4622-4. Epub 2018 Aug 8. PMID 30091121